CLINICAL TRIAL: NCT06236854
Title: Investigating the Link Between Preoperative Glymphatic Transport and Postoperative Delirium
Brief Title: Neuroimaging Risk of Postoperative Delirium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: NeuRO-POD
Record Dates: First submitted 2023-10-10; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-10

CONDITIONS: Post-operative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD-Absent: The group of older-aged surgical patients who are not diagnosed with delirium as assessed for the following fives days post-surgery.
  Interventions: Other: Delirium assessment (observational, not interventional)
- POD-Present: The group of older-aged surgical patients who are diagnosed with delirium as assessed for the following fives days post-surgery.
  Interventions: Other: Delirium assessment (observational, not interventional)

INTERVENTIONS:
Other: Delirium assessment (observational, not interventional) — As an observational study, we will assess the presence of postoperative delirium in the enrolled patients, which will define their group membership.

SUMMARY:
Postoperative delirium (POD) is a frequent disorder of consciousness, arousal and attention in elderly patients following surgery. The glymphatic system is a newly discovered waste cleaning system of the brain. Glymphatic transport of CSF has been shown to be impaired by perioperative factors. Reduced glymphatic transport has been related to a vicious cycle of neuroinflammatory marker build-up, leading to increased glymphatic transport impairment, leading eventually to neuronal damage and hence cognitive impairment. Therefore, glymphatic transport impairment has been suggested to be an important mechanism underlying POD. But not everyone who undergoes surgery presents POD, so what makes certain patients susceptible to POD? It has been suggested that glymphatic transport may already be impaired at preoperative baseline, which, with the added burden of perioperative strain on the system, 'tilts' the patient into POD. The primary aim of the current study is to measure glymphatic transport in patients preoperatively and assess whether patients who present POD ('POD patients') show impairments in preoperative glymphatic transport, relative to patients who do not present POD ('noPOD patients'). Two aspects of glymphatic transport will be assessed using two noninvasive MR techniques - fast-acquisition BOLD-fMRI and DTI-MR. POD will be assessed using the 3D-CAM questionnaire and patients will also be assessed preoperatively for symptoms of depression, state/trait anxiety and cognitive status using standardised self-report measures.

DETAILED DESCRIPTION:
Delirium is a fluctuating disturbance of consciousness with accompanying impairments in attention, cognition, perception, emotional regulation, psychomotor abilities as well as sleep-wake cycle regulation. Delirium frequently occurs following surgery with general anaesthesia and presents a common postoperative complication in elderly patients (>=65 years). 'Postoperative delirium' (POD) refers to the occurrence of delirium from as early as the timepoint immediately following surgery, i.e., at emergence from general anaesthesia, and up to 30 days following surgery. The reported occurrence of POD is highly variable, ranging from 10% to 70%, depending on the age of patients, diagnostic criteria, and the type of surgery. Those especially vulnerable are the oldest patients with the most medically complex cases undergoing cardiac, vascular, or hip fracture surgery. POD is associated with functional decline; a linear association between mortality and number of delirious days has been reported. POD has also been shown to increase risk of dementia up to 10-fold alongside a 2-fold increase in risk of institutionalisation and death. POD increases the length of general hospital stay and is associated with more than doubling one-year medical costs. Hence, there is a drive to elucidate the mechanisms of POD and identify risk factors that can facilitate adequate patient care management to reduce POD occurrence, both from a health and a costs perspective.

Several risk factors for POD have been identified, which can be categorised into two groups based on when they occur relative to surgery. Preoperative 'baseline' risk factors for POD include older age, pre-existing cognitive impairment, sensory and functional impairment, use of psychotropic drugs, history of major depressive disorder (MDD), institutional residence and greater comorbidity, especially with regards to cardiovascular disease. Peri-/intraoperative 'precipitating' risk factors include perioperative pain, environmental unfamiliarity, type of surgery, disrupted sleep, anaesthetic dosage, use of a bladder catheter and the type of medications used. An individual's risk of POD has been modelled as a sum of these baseline and precipitating risk factors, where a heightened burden of baseline preoperative factors necessitates fewer peri/intraoperative precipitating factors to induce POD. This interaction between baseline and precipitating factors follows the hypothesis of neural functional reserve, which suggests that an individual's ability to tolerate situations that encompass stress to the brain or brain 'injury' is dependent upon their baseline functional reserve - representing a patient's 'resilience'. Baseline preoperative risk factors of POD can be seen as factors that reduce a patient's reserve or resilience, and peri-/intraoperative 'precipitating' risk factors can be seen as prime examples of situations encompassing stress on the brain. A low functional reserve has been shown to be an independent risk factor for POD. Therefore, investigations of the underlying baseline preoperative neurological impairments that have the effect of reducing a patient's resilience to peri-/intraoperative stressors - and increase their risk of POD - are highly warranted. The investigators will assess whether two potential baseline preoperative neural impairments contribute to a patient's risk of POD.

The glymphatic system is a recently discovered waste clearance system of the brain, utilising the perivascular channels to sweep cerebrospinal fluid (CSF) through and away from the brain's parenchyma, taking waste products and extracellular metabolites with it, essentially cleaning the brain. Aquaporin-4 water channels located at astrocytic end-feed form an essential component of this system, facilitating CSF movement from perivascular spaces into the interstitial space. There are a small number of non-invasive measures available to assess aspects of glymphatic system function in humans. The first measure was proposed by whereby fast fMRI acquisition (TR<400ms) - with the boundary edge of the volume (i.e., slice 0) placed at the level of the fourth ventricle - allows for the detection of fluid inflow arriving at the edge of the imaging volume with high signal intensity. The acquired CSF signal with slow oscillations at around 0.05Hz were found to be of significantly higher amplitude during sleep vs. wake, driven by slow neural oscillations in the delta range (~1-4Hz), and was anticorrelated with fluctuations in the global grey matter BOLD signal. A decrease in this anticorrelation was reported in patients with Parkinson's disease and was significantly related to lower cognitive performance on the Montreal Cognitive Assessment tool. A relationship between reduced global BOLD-CSF flow coupling and severity of small vessel disease has been reported, related to increased dilation of the perivascular space. Hence, the global BOLD-CSF coupling could provide an indication as to impaired glymphatic transport.

A second recent approach was developed using diffusion tensor imaging (DTI) of diffusion-weighted images to evaluate the motion of water molecules along deep medullary veins and their accompanying perivascular spaces running perpendicular to the ventricular walls on a transverse slice at the level of the lateral ventricle bodies. At this location, the distribution of different fibre types allows for the discernment of water diffusivity along the perivascular space independently from that within corticofugal corona radiata projection fibres (running in the craniocaudal direction, i.e., z-axis) and superior longitudinal fascicle association fibres (running in the anterior-posterior direction, i.e., y-axis). This approach, called the 'DTI-ALPS' method, i.e., 'diffusion tensor imaging along the perivascular space', can non-invasively measure glymphatic transport (i.e., CSF flow through the perivascular space) at this specific location, as the perivascular space runs perpendicular to both the projection and association fibres. Regions of interest are first manually labelled from a T1-weighted scan to measure diffusivities within these fibres along three directions (x, y, and z). Perivascular diffusion can be evaluated independently from diffusion along projection and association areas by identifying the ratio of the mean x-axis diffusivity in both areas to the mean diffusivity of these areas at the axes perpendicular to the x-axis and fibre tracts, i.e., the y-axis for projection fibres and z-axis for association fibres.

Perioperative factors such as the type of GA, in combination with various other perioperative factors, may alter postoperative brain function by affecting the glymphatic system. Dysfunction of this system that removes harmful metabolites from the brain can lead to neurological disorders and neuroinflammation. Reduced glymphatic system transport leads to an increased accumulation of amyloid-beta and tau, inducing neuroinflammation leading to a chain of processes that end in neuronal damage. Postoperative increases in amyloid-beta and tau have been reported and shown to be a risk factor for POD. As outlined above, different anaesthetics have differential effects on the glymphatic system, and anaesthetic type has been shown to be a risk factor for POD in patients. Volatile anaesthetics such as isoflurane or sevoflurane have a higher chance of causing POD, whereas intravenous anaesthetics such as dexmedetomidine and propofol seemingly rather have a protective effect against POD.

Elderly patients but not young people are highly susceptible to POD, triggering the question of why this group is selectively susceptible. As outlined previously, preoperative risk factors for POD include preclinical Alzheimer's disease, cerebral microemboli, vascular dementia, hyperglycaemia and other neurovascular diseases or neurodegeneration, all of which show glymphatic transport impairment. Ageing is associated with degenerative changes such as depolarised or downregulated aquaporin-4, sleep deprivation, and reduced cerebrovascular pulsatility, all of which have the potential to impair glymphatic system transport. In line with the functional reserve hypothesis, it has been suggested that susceptible patients at risk of POD have pre-existing glymphatic system impairment that progresses slowly without significant cognitive impairment, and that the perioperative risk factors exacerbate the pre-existing glymphatic damage beyond the compensatory limit, resulting in significant cognitive changes. This theory suggests that baseline preoperative measures of glymphatic system transport can be informative on the risk of POD. Our primary aim is to investigate whether baseline preoperative measures of glymphatic system transport can be useful in identifying patients at risk of POD, utilising the two non-invasive MR-based measures outlined previously.

The overall aim of the current study is to investigate potential underlying pathobiological mechanisms that contribute to POD, to further understand the mechanisms of this frequent disorder in the elderly and enhance perioperative care and patient management. Whether an impairment in glymphatic system transport at preoperative baseline can be informative on risk of POD will be assessed. All target values will be assessed at preoperative baseline. Assessment of whether a patient is classified as a 'POD patient' or a 'noPOD patient' is based on a diagnosis of delirium on any of the five days following surgery (including the day of surgery).

ELIGIBILITY:
Inclusion Criteria:

* >= 65 years of age
* Fluent in German
* Presence of at least one further risk factor for POD

Exclusion Criteria:

* Individuals who do not meet all inclusion criteria
* Scheduled for neurological surgery
* Pre-existing neurological structural impairments or previous brain surgery
* ASA status 4
* Contraindication to MRI (e.g., pacemakers, artificial heart valves, cardioseal, aneurysm clips, implanted magnetic metal parts (screws, plates from surgery), cochlear implants, metal splitters/grenade splinters, acupuncture needle, insulin pump, piercings that cannot be removed, etc)
* Scheduled for emergency procedures
* Subjects with fear of confined spaces

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Older-aged elective surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Component of the brain waste clearance system as measured via magnetic resonance imaging | Morning prior to surgery during 30 minute MR protocol
  Glymphatic system transport measured via diffusion tensor imaging/functional magnetic resonance imaging parameter of CSF flow coupling with global neurovascular activity at preoperative baseline is changed in POD-Present patients as compared with POD-Absent patients

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schneider, Prof, Study Chair — Klinikum rechts der Isar der Technischen Universität München
Locations (1):
- Klinikum rechts der Isar der Technischen Universität München, München, Bavaria, Germany

REFERENCES:
- [Background] Fultz NE, Bonmassar G, Setsompop K, Stickgold RA, Rosen BR, Polimeni JR, Lewis LD. Coupled electrophysiological, hemodynamic, and cerebrospinal fluid oscillations in human sleep. Science. 2019 Nov 1;366(6465):628-631. doi: 10.1126/science.aax5440. PMID 31672896
- [Background] Taoka T, Masutani Y, Kawai H, Nakane T, Matsuoka K, Yasuno F, Kishimoto T, Naganawa S. Evaluation of glymphatic system activity with the diffusion MR technique: diffusion tensor image analysis along the perivascular space (DTI-ALPS) in Alzheimer's disease cases. Jpn J Radiol. 2017 Apr;35(4):172-178. doi: 10.1007/s11604-017-0617-z. Epub 2017 Feb 14. PMID 28197821
- [Background] Ren X, Liu S, Lian C, Li H, Li K, Li L, Zhao G. Dysfunction of the Glymphatic System as a Potential Mechanism of Perioperative Neurocognitive Disorders. Front Aging Neurosci. 2021 Jun 7;13:659457. doi: 10.3389/fnagi.2021.659457. eCollection 2021. PMID 34163349
- [Background] Han F, Chen J, Belkin-Rosen A, Gu Y, Luo L, Buxton OM, Liu X; Alzheimer's Disease Neuroimaging Initiative. Reduced coupling between cerebrospinal fluid flow and global brain activity is linked to Alzheimer disease-related pathology. PLoS Biol. 2021 Jun 1;19(6):e3001233. doi: 10.1371/journal.pbio.3001233. eCollection 2021 Jun. PMID 34061820
- [Background] Han F, Brown GL, Zhu Y, Belkin-Rosen AE, Lewis MM, Du G, Gu Y, Eslinger PJ, Mailman RB, Huang X, Liu X. Decoupling of Global Brain Activity and Cerebrospinal Fluid Flow in Parkinson's Disease Cognitive Decline. Mov Disord. 2021 Sep;36(9):2066-2076. doi: 10.1002/mds.28643. Epub 2021 May 17. PMID 33998068